CLINICAL TRIAL: NCT00274963
Title: Treatment of Relapsed / Refractory Chronic Lymphocytic Leukemia (CLL) WITH Bendamustine / Mitoxantrone (BM)
Brief Title: Bendamustine and Mitoxantrone in Treating Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: CLL2K; EU-20551; RIBOSEPHARM-GCLLSK-CLL2K
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: B-cell chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bendamustine Hydrochloride; Mitoxantrone

INTERVENTIONS:
Drug: bendamustine hydrochloride
Drug: mitoxantrone hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as bendamustine and mitoxantrone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving bendamustine together with mitoxantrone works in treating patients with relapsed or refractory B-cell chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate (remission rate) in patients with relapsed or refractory B-cell chronic lymphocytic leukemia (CLL) treated with bendamustine and mitoxantrone hydrochloride.

Secondary

* Determine the progression-free survival and overall survival of patients treated with this regimen.
* Determine the safety and tolerability of this regimen in these patients.

OUTLINE: This is a non-randomized, multicenter study.

Patients receive bendamustine IV over 1 hour on days1-3 and mitoxantrone hydrochloride IV over 30 minutes on day 1. Treatment repeats every 28 days for at least 2 courses in the absence of disease progression or unacceptable toxicity. Patients with responding disease (i.e., complete response or partial response) after 2 courses receive 2 additional courses of treatment for a total of 4 courses.

After completion of study treatment, patients are followed periodically for survival.

PROJECTED ACCRUAL: A total 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cytologically and immunophenotypically confirmed diagnosis of B-cell chronic lymphocytic leukemia (CLL)

  * Relapsed or refractory disease

PATIENT CHARACTERISTICS:

* No known hypersensitivity to any of the study medications
* No uncontrolled infection
* No impaired organ function

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2004-10; Primary Completion 2007-11 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Overall remission rate (partial and complete remission)

SECONDARY OUTCOMES:
Time to progression
Safety and tolerability
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Koeppler, MD, Study Chair — Praxis fuer Haematologie und Onkologie
Locations (12):
- Germany (12):
  - Humaine - Clinic, Bad Saarow
  - Schwerpunktpraxis fuer Haematologie und Internistische Onkologie, Berlin
  - Praxis Fuer Haematologie Internistische Onkologie, Cologne
  - Internistische Gemeinschaftspraxis - Halle, Halle
  - St. Marien Hospital, Hamm
  - Praxis fuer Haematologie und Onkologie, Koblenz
  - Haematologische / Onkologische Schwerpunktpraxis, Krefeld
  - Internistische Onkologische Praxis - Kronach, Kronach
  - Internistische Praxis - Neuss, Neuss
  - Internistische Gemeinschaftspraxis - Oldenburg, Oldenburg
  - Haematologische Praxis, Weiden
  - Deutsche Klinik fuer Diagnostik, Wiesbaden

REFERENCES:
- [Result] Koppler H, Fuss H, Hurtz HJ, Knigge O, Losem C, Reschke D, Schmitz S, Weide R, Weiss J, Hallek M; GCLLSG. Bendamustine plus mitoxantrone for relapsed/refractory chronic lymphocytic leukaemia (CLL): results of a multicentre phase II study of the German CLL Study Group (GCLLSG). Br J Haematol. 2012 Jul;158(2):238-241. doi: 10.1111/j.1365-2141.2012.09132.x. Epub 2012 May 10. PMID 22571691